CLINICAL TRIAL: NCT03416738
Title: (C-STAR) Center for the Study of Aphasia Recovery Modeling Treated Recovery From Aphasia
Brief Title: Modeling Treated Recovery From Aphasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Julius Fridriksson, Endowed Professor, University of South Carolina
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00053559; P50DC014664 (NIH)
Record Dates: First submitted 2018-01-23; First posted 2018-01-31 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Aphasia; Stroke; Stroke, Ischemic; Aphasia, Broca; Aphasia, Global; Aphasia, Mixed; Aphasia, Jargon; Aphasia, Expressive; Aphasia, Conduction; Aphasia, Fluent; Aphasia, Anomic
MeSH Terms: conditions — Aphasia; Stroke; Ischemic Stroke; Aphasia, Broca; Aphasia, Wernicke; Aphasia, Conduction; Anomia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Semantically focused treatment (Active Comparator): This treatment will focus on improving word finding and comprehension of information.
  Interventions: Behavioral: Semantically focused treatment
- Phonologically focused treatment (Active Comparator): This treatment will focus on training speech sound production, targeting overall production abilities.
  Interventions: Behavioral: Phonologically focused treatment

INTERVENTIONS:
Behavioral: Semantically focused treatment — Tasks are as follows:
  1. Semantic feature analysis (SFA): For each pictured stimulus the patient is prompted to name the picture, and then to produce related words that represent features similar to the target word.
  2. Semantic barrier task: The goal is for one participant (e.g., patient) to describe each card so that the other participant (e.g., clinician) can guess the picture on the card. Participants are only allowed to describe the semantic features of the target and the clinician models the kinds of cues that are allowed.
  3. Verb network strengthening treatment (VNeST): This treatment targets lexical retrieval of verbs and their thematic nouns. The objective of VNeST is for the patient to generate verb-noun associates with the purpose of strengthening the connections between the verb and its uses.
  These are tasks used in clinical aphasia rehabilitation.
  Arms: Semantically focused treatment
Behavioral: Phonologically focused treatment — Tasks are as follows:
  1. Phonological (sound) components analysis task: Participants are to name a given picture and then to identify the sound features of the target words (e.g., first sound, last sound, and rhyme).
  2. Phonological production task: This tasks asks participants to sort and identify the sounds that make up a word. Various stages include identifying first sounds, last sounds, etc. Participants also work on blending sounds together to form words.
  3. The phonological judgment task: A computerized presentation of verbs and nouns where participants are required to judge whether pairs of words include similar phonological features.
  These are tasks used in clinical aphasia rehabilitation.
  Arms: Phonologically focused treatment

SUMMARY:
Stroke is the leading cause of adult disability in the United States, and aphasia is common following a stroke to the left hemisphere of the brain. Aphasia therapy can improve aphasia recover; however, very little is known about how different patients respond to different types of treatments.

The purpose of this study is to understand how the following factors influence an individual's response to aphasia treatment: 1) biographical factors (e.g., age, education, gender), 2) post-stroke cognitive/linguistic abilities and learning potential, and 3) the location and extent of post-stroke brain damage. We are also interested in understanding the kinds of treatment materials that should be emphasized in speech/language treatment.

Overall, the goal of the current research is to inform the clinical management of post-stroke aphasia by identifying factors that can predict how an individual will respond to different treatment methods.

ELIGIBILITY:
Inclusion Criteria:

* Experienced a left hemisphere ischemic or hemorrhagic stroke At least 12 months post-stroke
* Primarily English speaker for the past 20 years
* Ability to provide informed written or verbal consent MRI-compatible (e.g., no metal implants, not claustrophobic)

Exclusion Criteria:

* History of a right hemisphere stroke (Bilateral stroke)
* Clinically reported history of dementia, alcohol abuse, psychiatric disorder, traumatic brain injury, or extensive visual acuity or visual-spatial problems
* Severely limited speech production and/or auditory comprehension that interferes with adequate participation in the therapy provided

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2016-08-02 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Philadelphia Naming Test | 6 months
  Assesses the ability to name functional objects

CONTACTS AND LOCATIONS:
Overall Officials: Julius Fridriksson, PhD, CCC-SLP, Principal Investigator — University of South Carolina
Locations (2):
- United States (2):
  - Medical University of South Carolina, Charleston, South Carolina
  - University of South Carolina, Columbia, South Carolina

REFERENCES:
- [Derived] Busby N, Wilmskoetter J, Gleichgerrcht E, Rorden C, Roth R, Newman-Norlund R, Hillis AE, Keller SS, de Bezenac C, Kristinsson S, Fridriksson J, Bonilha L. Advanced Brain Age and Chronic Poststroke Aphasia Severity. Neurology. 2023 Mar 14;100(11):e1166-e1176. doi: 10.1212/WNL.0000000000201693. Epub 2022 Dec 16. PMID 36526425
- See also: Study website — https://cstar.sc.edu

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-20): https://cdn.clinicaltrials.gov/large-docs/38/NCT03416738/Prot_SAP_001.pdf